CLINICAL TRIAL: NCT01231295
Title: Evaluating the Performance of Isotopic Brain Imaging of Glucose Metabolism Via PET (18F-FDG) and Perfusion SPECT (99mTc-ECD) for the Diagnosis of Prodromal Stage Alzheimer's Disease
Brief Title: Isotopic Imaging for Prodromal Alzheimer's Disease
Acronym: ISALP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-N/2009/POK-01; 2009-013476-53 (EudraCT Number)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 x 10ml of blood and 3 ml lumbar puncture for Abeta1-40, A1beta-42, Abetan-40, Abetan-42, sAPPalpha, Tau, pTau, and DNA extraction for the ApoE4 gene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Memory problems: Group with clinically validated memory problems
- Reference group: Group without memory problems

SUMMARY:
The primary objective of this study is to characterize cerebral metabolism modifications using 18F-FDG PET technology and perfusion with 99MTC-ECD SPECT in patients with prodromal Alzheimer's Disease drawn from a high risk population. We also compare PET and SPECT imaging within this framework, and search for optimal diagnostic thresholds.

ELIGIBILITY:
Inclusion Criteria for the group with memory problems:

* patient consulting for memory problems
* caucasian
* memory complaint is validated by a clinical evaluation
* cognitive performance is sufficiently well preserved so that a diagnostic of dementia cannot be made (according to the DSM-IV-R and NINCDS-ADRDA criteria) at the time of inclusion
* the patient speaks French
* presence of an informant
* accepts to sign consent

Inclusion Criteria for the group without memory problems (reference population):

* at least four years of formal education
* patient consulting for memory problems
* memory problem reported by the patient is not validated by the consultation, nor by the battery of tests specified during screening
* presence of an informant
* Clinical Dementia Rating (CDR) = 0
* accepts to sign consent

Exclusion Criteria:

* Instrumental Activities of Daily Living (IADL): at least two items > 1
* Anticholinesterasic treatments and/or memantin before study inclusion
* major depressive syndrome, according to the Global Depressive Scale
* Known neurodegenerative disease or general disease or major physical problems that could interfere with cognitive functioning and testing
* Pathology that might lead to death in the short term (evolving cancer, non stable cardiopathy, hepatic, renal or respiratory insufficiency)
* contra-indications for MRI, PET or SPECT scans
* not affiliated with a social security regimen

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of elderly patients over 70 years of age who consult for memory problems. These patients are further split into two groups based on the clinical validation of memory complaints.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2011-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The difference between AUCs for PET and SPECT imaging | 1 month
  The difference between the AUCs (area under the curve) for PET and SPECT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Olivier Kotzki, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (25):
- France (25):
  - CHU d'Amiens - Hôpital Sud, Amiens
  - CHU d'Angers - Hôtel-Dieu, Angers
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - APHP - Hôpital Albert Chenevier, Créteil
  - APHP - Hôpital Charles Foix, Ivry-sur-Seine
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - APHP - Hôpital Emile Roux, Limeil-Brévannes
  - APHM - Hôpital La Timone Adultes, Marseille
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nancy - Hôpital Central, Nancy
  - CHU de Nice - Hôpitaux L'Archet 1 et 2, Nice
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - APHP - Hôpital Lariboisière, Paris
  - APHP - Hôpital Broca, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims - Hôpital Maison Blanche, Reims
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHRU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHRU de Toulouse - Hôpital Garonne, Toulouse
  - CHRU de Toulouse - Hôpital Purpan, Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours